CLINICAL TRIAL: NCT00954655
Title: Genetic Risk Factors for Gastrointestinal Stromal Tumors (GIST)
Brief Title: Study of Tumor Samples in Patients Undergoing Treatment for Gastrointestinal Stromal Tumors on Clinical Trial ACOSOG-Z9001
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z9081; ACOSOG-Z9081; CDR0000631512 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1: Tumor samples are used for polymorphism and mutation analysis.
  Interventions: Genetic: mutation analysis; Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor samples in patients undergoing treatment for gastrointestinal stromal tumors on clinical trial ACOSOG-Z9001.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine polymorphisms in selected genes involved in the detoxifying/metabolizing and DNA repair pathways in relation to specific mutations and types of mutation in the c-kit gene in tumor tissue from patients with gastrointestinal tumors (GIST) undergoing treatment on clinical trial ACOSOG-Z9001.

Secondary

* To examine approximately 758 polymorphisms among candidate genes involved in detoxification/metabolism, cell cycle control, and DNA damage/repair in relation to specific mutations and types of mutation in the c-kit gene in tumor tissue from GIST patients for hypothesis generation. (exploratory)
* To conduct an exploratory analysis of the polymorphism distribution in these patients. (exploratory)
* To examine the association between the above polymorphisms and major toxicity (Grade 3/4) of adjuvant imatinib mesylate. (exploratory)

OUTLINE: Tumor samples are used for polymorphism and mutation analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor samples from patients with gastrointestinal stromal tumors enrolled on clinical trial ACOSOG-Z9001

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumor samples from patients with gastrointestinal stromal tumors enrolled on clinical trial ACOSOG-Z9001
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Engel, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States